CLINICAL TRIAL: NCT06770725
Title: Investigating the Effect of the Temporal Adaptation Approach on Activity Self-Efficacy, Time Perception, and Daily Activity Routine With Executive Skills in Children With ADHD: A 1-Month Follow-Up Randomized Controlled Study
Brief Title: Investigating the Effects of the Temporal Adaptation Approach in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gonca Bumin, Supervisor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61351342 / ARALIK 2023-06
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Temporal Adaptation; Time Management; Time Perception; Occupational self-efficacy; Executive Functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The participants who are allocated to the Control Group arm will receive conventional occupational therapy interventions for the duration of the study.
  Interventions: Behavioral: Conventional Occupational Therapy
- Experimental Group (Experimental): Participants allocated to the Experimental Group will receive Temporal Adaptation Intervention during the study.
  Interventions: Behavioral: Temporal Adaptation Intervention

INTERVENTIONS:
Behavioral: Temporal Adaptation Intervention — The research on temporal adaptation intervention will be conducted through activities and individual sessions within the framework of temporal adaptation intervention. The activities included in the temporal adaptation intervention used in our research have been adapted for ADHD by referencing temporal adaptation training models in the literature.
  Arms: Experimental Group
Behavioral: Conventional Occupational Therapy — The control group will be given a 10-week-long conventional occupational therapy intervention by the investigator (Fatma Temizkan). The intervention will consist of occupational therapy approaches such as; obstacle courses, sensory integration, motor skills training, cognitive skills training, sequenced activities and so on.
  Arms: Control Group

SUMMARY:
This study investigates the impact of temporal adaptation interventions on children with Attention Deficit Hyperactivity Disorder (ADHD), focusing on activity self-efficacy, time perception, daily activity routines, and executive functions. The intervention aims to address the challenges ADHD children face in time processing abilities, which include understanding the concept of time, being punctual, initiating and completing daily activities independently, planning and completing long-term projects, using a calendar, and hurrying when necessary.

The research will be conducted at the Hacettepe University Faculty of Health Sciences Department of Occupational Therapy's educational and research units. Participants will be children diagnosed with ADHD by a Child and Adolescent Psychiatrist. These children will then be randomly assigned to control and training groups. A total of 60 individuals, 30 for each group, will be included in the study based on power analysis. The effectiveness of the study will be shared, and should it prove effective, the same study will be replicated with the control group.

The intervention consists of activities designed to enhance temporal adaptation, adapted for ADHD from models in the literature. Over 10 weeks, the children will engage in weekly 60-minute sessions, each week focusing on different activities to improve temporal adaptation skills. Activities include teaching concepts of calendars and clocks, rhythm exercises with metronomes, time estimation games, daily and weekly planner preparation, time matching games, and exercises to improve time management and planning abilities.

Data will be collected using various tools including a demographic information form, time perception threshold measurement tasks, temporal production tasks, Child Activity Self-Assessment Scale (COSA), and Executive Functions and Occupational Routines Scale (EFORTS). The study's hypotheses test the null hypothesis that temporal adaptation intervention does not affect activity self-efficacy, time perception, daily activity routine, and executive functions in children aged 9-12 with ADHD.

This comprehensive approach aims to enhance the daily lives of children with ADHD by improving their ability to manage time effectively, thereby positively affecting their education, self-care, social relationships, and overall quality of life.

DETAILED DESCRIPTION:
This study explores the efficacy of a temporal adaptation intervention in enhancing the quality of life and functional abilities of children diagnosed with Attention Deficit Hyperactivity Disorder (ADHD). ADHD is a neurodevelopmental disorder characterized by patterns of inattention, impulsivity, and hyperactivity that detrimentally influence an individual's academic, social, motor, sensory, and executive functioning. Notably, children with ADHD often struggle with time processing abilities, which can manifest as difficulties in understanding time concepts, adhering to schedules, and managing daily activities.

Background ADHD significantly impacts the cognitive and behavioural domains of affected children, leading to challenges in daily living and academic achievement. Previous research has identified specific issues in time perception and temporal processing among children with ADHD, including time duration discrimination and time reproduction. These difficulties extend to both the understanding and management of time, impacting their daily routines and task completion. Functional and structural imaging studies have shown that the brain regions involved in time processing overlap with areas implicated in the pathogenesis of ADHD, such as the neocerebellum, basal ganglia, and prefrontal cortex. Given the centrality of time management skills to academic performance, self-care, and social interactions, interventions aimed at improving these skills could significantly enhance the functional outcomes for children with ADHD.

Objective The primary objective of this research is to evaluate the effectiveness of a temporal adaptation intervention aimed at improving activity self-efficacy, time perception, daily activity routines, and executive functions among children with ADHD. The intervention seeks to address the specific temporal processing challenges faced by these children, potentially leading to better time management, planning, and organizational skills.

Methods The intervention will be structured around a series of activities and individual sessions designed based on models of temporal adaptation training adapted for ADHD. These activities will target the development of skills related to the understanding and management of time, such as using calendars and clocks, estimating the duration of activities, and planning and executing daily and long-term tasks.

Setting and Participants The research will be carried out at a university's health sciences faculty, utilizing its educational and research facilities. The study will include children who meet the inclusion criteria of being diagnosed with ADHD, within the age range of 9-12 years, and voluntarily agree to participate. Exclusion criteria include the presence of additional diagnoses and the unwillingness of parents to adhere to the intervention protocols.

Design A randomized controlled trial design will be employed, with participants being randomly assigned to either the intervention or control group. The intervention group will undergo the temporal adaptation training program, while the control group will receive no such training. The training program will span 10 weeks, with sessions held once a week for 60 minutes. Each session will focus on different activities tailored to improve temporal adaptation, such as teaching time concepts, rhythm exercises with a metronome, and games designed to enhance time estimation and planning skills.

Assessment Tools

A comprehensive set of tools will be used to evaluate the impact of the intervention on the participants, including:

Demographic Information Form: To collect baseline demographic data. Time Perception Threshold Measurement: To assess the ability to discriminate between different durations.

Temporal Production Task: To evaluate the accuracy of reproducing time intervals.

Child Activity Self-Assessment Scale (COSA): To measure perceived efficacy and importance in daily activities.

Executive Functions and Occupational Routines Scale (EFORTS): To assess executive functioning and daily routines.

Hypotheses The study will test several hypotheses, including the assumption that the temporal adaptation intervention has no effect on the measured outcomes. The alternative hypothesis posits that the intervention will significantly improve activity self-efficacy, time perception, daily activity routines, and executive functions in participating children.

Data Analysis Statistical analyses will be conducted using appropriate software, with comparisons made between pre- and post-intervention assessments within and between the intervention and control groups. The effectiveness of the intervention will be determined through Cohen's Effect Size, with predefined criteria for interpreting the magnitude of the effect.

Conclusion This study aims to provide evidence on the effectiveness of a temporal adaptation intervention for children with ADHD, focusing on enhancing their ability to understand and manage time. By improving time management and planning skills, the intervention seeks to positively affect educational achievements, self-care, social relationships, and overall quality of life for these children.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 9 and 12 years of age.
* Clinical diagnosis of Attention Deficit Hyperactivity Disorder (ADHD)
* Must be willing to participate and adhere to the study protocols

Exclusion Criteria:

* Additional psychiatric or developmental diagnoses that can interfere with the study outcomes

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Time Perception Threshold Measurement | From enrollment to the end of treatment at 10 weeks
  Assesses the ability to discriminate between different durations.
Temporal Production Task | From enrollment to the end of treatment at 10 weeks
  Evaluates the accuracy of reproducing time intervals.
Child Occupational Self-Assessment Scale | From enrollment to the end of treatment at 10 weeks
  The Child Occupational Self-Assessment Scale measures perceived efficacy and importance in daily activities. The scale consists of 25 items that evaluate the children's perceived occupational performance and the importance of the occupations under seven areas. All questions are scored from 1 to 4. The scale yields 14 different sub-scores (a performance and an importance score for each area). The Communication and the Executive Functions sub-scores range between 6 and 24, the Motor Skills sub-scores range between 3 and 12, the Academic sub-scores range between 5 and 20 and the Self Regulation, Intrumental Activities of Daily Living and Activities of Daily Living sub-scores range between 2 and 8. For the performance sub-scores, a higher score indicate better perceived performance. For the importance sub-scores, a higher score indicate higher given importance.
Executive Functions and Occupational Routines Scale | From enrollment to the end of treatment at 10 weeks
  The scale ssesses executive functioning and daily routines. The scale consists of 30 items, divided into subscales based on everyday functional routines, scored from 1 (never) to 5 (always). The scale does not have a total score, rather, a mean score is calculated for each sub-scale as well as the total scale. The mean score ranges between 1 and 5, with with higher scores indicating better executive control.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, PhD., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that are collected in this study contain individuals' performance scores on various tests, which can be indirectly related to their academic success and overall academic performance. Therefore, the informed consent that is collected from the participants states that their data will not be shared with third parties (any person or institution except for the research team and related ethical boards) except for ethical committees. Therefore, the data will not be shared with other researchers.